CLINICAL TRIAL: NCT06993818
Title: Evaluatıon Of Asprosın And Tumor Necrosıs Factor-α Levels In Gıngıval Crevıcular Fluıd And Serum Of Patıents Wıth Controlled And Uncontrolled Type 2 Dıabetıc Chronic Periodontitis
Brief Title: Asprosın And Tumor Necrosıs Factor-α Levels In Type 2 Dıabetıc Chronıc Periodontitis
Status: Completed | Type: Observational
Sponsor: Eda Cetin Ozdemir (Other)
Responsible Party: Sponsor-Investigator, Eda Cetin Ozdemir, Principal Investigator, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Other Study IDs: Kahramanmaraş Sütçü İmam Unive
Record Dates: First submitted 2025-05-13; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis; Diabetes Mellitus; Asprosin levels
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control Group: systemically and periodontally healthy control group: Periodontal clinical parameters and examination of asprosin levels in gingival crevicular fluid and serum samples
  Interventions: Other: Gingival Crevicular Fluid; Diagnostic Test: Serum Asprosin
- Uncontrolled T2DM-CP: Stage III Grade C Periodontitis, Uncontrolled T2DM group: Periodontal clinical parameters and examination of asprosin levels in gingival crevicular fluid and serum samples
  Interventions: Other: Gingival Crevicular Fluid; Diagnostic Test: Serum Asprosin
- Controlled T2DM-CP: Stage III Grade B Periodontitis, Controlled T2DM: Periodontal clinical parameters and examination of asprosin levels in gingival crevicular fluid and serum samples
  Interventions: Other: Gingival Crevicular Fluid; Diagnostic Test: Serum Asprosin
- CP: Stage III Grade B Periodontitis group: Periodontal clinical parameters and examination of asprosin levels in gingival crevicular fluid and serum samples
  Interventions: Other: Gingival Crevicular Fluid; Diagnostic Test: Serum Asprosin

INTERVENTIONS:
Other: Gingival Crevicular Fluid — Periodontal clinical parameters and examination of asprosin levels in gingival crevicular fluid and serum samples
Diagnostic Test: Serum Asprosin — Periodontal clinical parameters and examination of asprosin levels in gingival crevicular fluid and serum samples

SUMMARY:
Periodontal disease is a chronic, multifactorial inflammatory disease in which biochemical and cellular events trigger each other, leading to the destruction of the tissues supporting the teeth . The pathogenesis of the disease is a dynamic process that develops as a result of complex interactions between pathogenic bacteria and the host response . There is a bidirectional relationship between diabetes mellitus (DM), which is among the systemic diseases that negatively affect the host immune response, and periodontal disease. In the case of DM, long-term hyperglycemia causes proteins to react irreversibly with glucose, resulting in the formation of advanced glycation end products (AGEs). It is suggested that increased AGE levels increase cytokine secretion against periodontopathogens, exacerbate inflammatory tissue destruction, and may negatively affect biological functions through cell-cell and cell-matrix interactions in the connective tissue.

The present study was conducted to gain further insight into the role of CGF and serum Asprosin level in the pathogenetic processes linking DM and periodontal disease.

DETAILED DESCRIPTION:
Periodontal disease is a chronic, multifactorial inflammatory disease in which biochemical and cellular events trigger each other, leading to the destruction of the tissues supporting the teeth . The pathogenesis of the disease is a dynamic process that develops as a result of complex interactions between pathogenic bacteria and the host response . There is a bidirectional relationship between diabetes mellitus (DM), which is among the systemic diseases that negatively affect the host immune response, and periodontal disease . In the case of DM, long-term hyperglycemia causes proteins to react irreversibly with glucose, resulting in the formation of advanced glycation end products (AGEs). It is suggested that increased AGE levels increase cytokine secretion against periodontopathogens, exacerbate inflammatory tissue destruction, and may negatively affect biological functions through cell-cell and cell-matrix interactions in the connective tissue . Periodontitis, a widespread infectious disease, is also considered a systemic inflammation. In the presence of periodontitis, some inflammatory cytokines are produced in periodontal tissues and their levels in the circulation also increase . It has been reported that the levels of Tumor necrosis factor-α (TNF-α), which is considered an acute phase reactant, are increased in the adipose tissue of diabetic rodents. TNF-α has proinflammatory properties and can reduce insulin sensitivity . Studies have shown that diabetic monocytes secrete 24-32 times more TNF-α; this situation is associated with the development and progression of diabetic periodontitis. Adipokines are important molecules secreted from adipose tissue and play a role in various physiological processes such as energy intake, blood pressure, metabolism and inflammation . In 2016, Romere et al. showed that plasma levels of Asprosin, encoded by the Fibrillin-1 gene, increase in the fasting state and decrease after meals. After crossing the blood-brain barrier, the asprosin hormone stimulates the orexigenic (appetite-increasing) AgRP neuron group through a cAMP-dependent pathway activity. Simultaneously, gamma aminobutyric acid-dependent proopiomelanocortin neurons are suppressed, thus increasing appetite, obesity, and ultimately body weight . Asprosin is associated with diseases such as diabetes mellitus, obesity, polycystic ovary syndrome, and cardiovascular diseases . Recent studies have shown that asprosin plays a role in the inflammatory responses of many cell types. Asprosin increases B cell-dependent inflammation by inducing hepatic glucose synthesis and also increases blood glucose levels by inhibiting insulin secretion . Many studies have shown that serum asprosin concentrations in patients with type 2 diabetes mellitus are systemically higher than in healthy controls . However, the authors did not find any studies in the literature evaluating asprosin levels in individuals with type 2 DM and chronic periodontitis. In light of the previous studies summarized above, the present study was conducted to gain more insight into the role of CGF and serum Asprosin levels in the pathogenetic processes linking DM and periodontal disease. This study is the first to examine Asprosin levels in gingival crevicular fluid (GCF) and serum of CP patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a volunteer

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients applying to Kahramanmaraş Sütçü İmam University, Faculty of Dentisrty, Department of Periodontology.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Changes in Asprosin Levels in GCF an Serum Samples in periodontal disease | 6 Mounth
  Investigators expect a statistically significant difference between controlled and uncontrolled T2DM and CP patients and healthy individuals in terms of serum and CGF Asprosin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I dont want to share

REFERENCES:
- See also: Related Info — https://www.frontiersin.org/journals/endocrinology/articles/10.3389/fendo.2020.00064/full